CLINICAL TRIAL: NCT04015908
Title: A Multimodal Analgesia Protocol Adapted for Ambulatory Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121505
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-05

CONDITIONS: Opioid Use
MeSH Terms: interventions — Celecoxib; Acetaminophen; Pregabalin; Oxycodone; oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- multi-modal (Experimental): 3 Different Non-opioid pain medication taken every 6 hours
  Celecoxib 100mg
  Acetaminophen 325mg
  Pregabalin 50 mg
  Plus, for breakthrough pain
  oxycodone 5-10 mg will be taken every 4 hours as needed for pain.
  Interventions: Drug: Celecoxib; Drug: Acetaminophen; Drug: Pregabalin; Drug: Oxycodone
- Control (Active Comparator): 7 day supply of Percocet (oxycodone 5mg/acetaminophen 325 mg) to be taken 1-2 by mouth every 4 hours as needed for pain.
  Interventions: Drug: Percocet

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 100mg
  Other Names: Celebrex
  Arms: multi-modal
Drug: Acetaminophen — Acetaminophen 325mg
  Other Names: Paracetamol
  Arms: multi-modal
Drug: Pregabalin — Pregabalin 50 mg
  Other Names: Lyrica
  Arms: multi-modal
Drug: Oxycodone — oxycodone 5-10 mg
  Other Names: Xtampza ER, Oxaydo, Roxicodone
  Arms: multi-modal
Drug: Percocet — Percocet (oxycodone 5mg/acetaminophen 325 mg)
  Other Names: Oxycodone / Paracetamol
  Arms: Control

SUMMARY:
The primary objective of this trial is to determine whether the combination of three non-opioid analgesics (multimodal analgesia) can significantly reduce or eliminate the need for opioids after ambulatory surgery.

A secondary objective would be to present credible data for insurance providers about the opioid sparing effect of these medications. This data may encourage insurance providers to support payment for short term use of certain analgesics that currently require prior authorization.

DETAILED DESCRIPTION:
Prescription opioids are associated with addiction and accidental overdose, yet they continue to be the most commonly prescribed analgesics after ambulatory surgery.

Multimodal analgesia is a promising alternative to opioids. It is based on the theory that a combination of more than one analgesic (with non-opioid mechanisms of action) can provide pain relief equal to or exceeding that of traditional opioids.

Multimodal analgesia is not associated with opioid related side effects such as respiratory depression, nausea, constipation, and itching.

Implementation of multi-modal analgesia in an ambulatory setting is challenging for a number of reasons.

First, patient compliance with multiple medications and complex dosing schedules is poor.

Second, misinformation still exists about the dosing of acetaminophen and NSAIDS (non-steroidal anti-inflammatory drugs). For example, many patients and health care providers believe that acetaminophen and NSAIDS cannot be taken concurrently. As a result, the additive analgesic effect of combining these drugs is not achieved.

Finally, some medications used for multimodal analgesia can be difficult to procure in the ambulatory setting. For example, pregabalin (trade name Lyrica) has been used successfully to treat acute pain and reduce opioid requirements after surgery. However, its mechanism of action is similar to that of gabapentin (an older and less expensive drug) and insurers are reluctant to approve its use over the expensive alternative.

Although gabapentin is a useful analgesic for chronic pain, its delayed onset of activity and unpredictable blood levels after oral administration make it impractical to use in the setting of acute pain. In fact, optimal dosing of gabapentin may require several days or weeks to establish.By contrast, pregabalin has a rapid onset of action with consistent and predictable plasma levels after oral administration.

For this trial, patients in the control group would receive traditional postoperative pain medication consisting of a combination of oxycodone and acetaminophen (trade name Percocet) as needed at 4-6 hour intervals.

Patients in the study group would receive the following:

* Three non-opioid pain medications (acetaminophen,celecoxib, and pregabalin) would be taken concurrently at six hour intervals for a period of 7 days.
* These three non-opioid medications (acetaminophen, celecoxib, and pregabalin ) would be provided in a "blister pack". All scheduled pain medication for a given 6 hour interval would be contained in a single compartment to simplify compliance for the patient. Study patients would also have access to oxycodone as a "rescue medication".

The principles of postoperative pain management addressed in this protocol are supported by existing literature.

1. Patient compliance with complex medication dosing protocols may be improved using calender and time based "blister packs".
2. Pain control using combined acetaminophen and NSAID is superior to that either drug in isolation
3. Pregabalin can reduce opioid requirements and opioid related nausea when treating acute pain.

The primary objective of this trial is to determine whether the combination of three non-opioid analgesics (multimodal analgesia) can significantly reduce or eliminate the need for opioids after ambulatory surgery.

A secondary objective would be to present credible data for insurance providers about the opioid sparing effect of these medications. This data may encourage insurance providers to support payment for short term use of certain analgesics that currently require prior authorization.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 18 and 65 having one of three elective procedures as an outpatient. These procedures are associated with moderate to severe postoperative pain (anterior cruciate ligament reconstruction (knee), ankle ligament reconstruction (foot/ankle), or ligament reconstruction with tendon interposition (hand))
* Patients should have operative risk category of American Society of Anesthesiologists (ASA) 1 or 2 .
* Patients weighing between 70-100kg will be included to allow standardization of medication dosing

Exclusion Criteria:

* Allergy to Study Medications
* Previous History of Chronic Opioid Use
* Patient Refusal to Participate
* Known of Suspected History of Sleep Apnea
* Known History of Chronic Pain Syndrome
* Weight less than 70kg or greater than 100kg due to standardization of medication doses.
* Revision Surgery
* Inability to take study medications due to medication incompatibility or co-existing disease
* Patients refusing or unable to receive US guided nerve block for postoperative pain
* Patients unable to read and comprehend written consent document

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Swenson, MS, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swenson JD, Conrad KM, Pace NL, Phillips K, Saltzman CL. Scheduled, Simultaneous Dosing of Pregabalin, Celecoxib, and Acetaminophen Markedly Reduces or Eliminates Opioid Use After ACL Reconstruction Using Allograft or Hamstring Tendon Autograft: A Randomized Clinical Trial. Orthop J Sports Med. 2022 Dec 8;10(12):23259671221140837. doi: 10.1177/23259671221140837. eCollection 2022 Dec. PMID 36518729

RESULTS

PARTICIPANT FLOW:
Groups:
- Multi-modal: 3 Different Non-opioid pain medication taken every 6 hours
  Celecoxib 100mg
  Acetaminophen 325mg
  Pregabalin 50 mg
  Plus, for breakthrough pain
  oxycodone 5-10 mg will be taken every 4 hours as needed for pain.
  Celecoxib: Celecoxib 100mg
  Acetaminophen: Acetaminophen 325mg
  Pregabalin: Pregabalin 50 mg
  Oxycodone: oxycodone 5-10 mg
Period: Overall Study
Arm/Group | Multi-modal | Control
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participant characteristics and anesthetics drugs
Groups:
- Total: Total of all reporting groups
Arm/Group | Multi-modal | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11) | 37 (11) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 13 | 18 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 169 (9) | 171 (8) | 170 (9)
Weight [Mean (Standard Deviation); unit: kg] | 75 (13) | 80 (13) | 76 (13)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26 (6) | 27 (4) | 27 (5)
Scopolamine patch [Count of Participants; unit: Participants] | 19 | 19 | 38
Intraoperative fentanyl [Mean (Standard Deviation); unit: mg] | 110 (45) | 110 (46) | 110 (45)
PACU fentanyl [Mean (Standard Deviation); unit: mg] | 93 (66) | 92 (77) | 93 (72)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Pain Experienced
Description: Pain as measured by a 0-10 Visual Analog Scale (VAS) pain scale, where "0" is the lowest score and "10" is the highest score. For example, 10 would be severe pain and 0 would be none. Cumulative scores were the total scores over 6 days and were expressed with the absolute totals with range. No subscales were used. Cumulative scores represent the absolute sum of each data point for 6 days. The total cumulative range for pain is 0-60.
Time Frame: Cumulative every day after 6 days post-operative
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Multi-modal | Control
Number analyzed (Participants) | 50 | 49
Score on a scale | 28 [14 to 35] | 35 [28 to 41]

2. Secondary Outcome: Amount of Nausea Experienced
Description: Nausea as measured by a 0-10 Visual Analog Scale (VAS) nausea scale, where "0" is the lowest score and "10" is the highest score. For example, 10 would be severe nausea and 0 would be none. Cumulative scores were the total scores over 6 days and were expressed with the absolute totals with range. No subscales were used. Cumulative scores represent the absolute sum of each data point for 6 days. The total cumulative range for nausea is 0-60.
Time Frame: Cumulative every day after 6 days post-operative
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Multi-modal | Control
Number analyzed (Participants) | 50 | 49
Score on a scale | 0 [0 to 0] | 0 [0 to 8]

3. Secondary Outcome: Amount of Itching Experienced
Description: Itching as measured by a 0-10 Visual Analog Scale (VAS) itching scale, where "0" is the lowest score and "10" is the highest score. For example, 10 would be severe itching and 0 would be none. Cumulative scores were the total scores over 6 days and were expressed with the absolute totals with range. No subscales were used. Cumulative scores represent the absolute sum of each data point for 6 days. The total cumulative range for itching is 0-60.
Time Frame: Cumulative every day after 6 days post-operative
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Multi-modal | Control
Number analyzed (Participants) | 50 | 49
Score on a scale | 0 [0 to 0] | 0 [0 to 4]

4. Secondary Outcome: Amount of Oxycodone Used
Description: Oxycodone use, measured by number of 5-mg tablets as standard dose
Time Frame: Cumulative every day after 6 days post-operative
Measure: Median (Inter-Quartile Range); unit: tablets
Arm/Group | Multi-modal | Control
Number analyzed (Participants) | 50 | 49
tablets | 0 [0 to 2] | 8 [1.25 to 16]

ADVERSE EVENTS:
Time Frame: 6 days
Arm/Group | Multi-modal | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

LIMITATIONS AND CAVEATS:
An important limitation of this trial is the inability to discern the true effects of medication delivery and medications received. This effect could only be measured by studying these 2 interventions separately. Similarly, this dosing regimen was applied to patients with a fixed range of weights and ages. The study design may have discouraged patients who prefer opioid analgesia. This could cause a sampling bias leading only patients motivated to use less opioid to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT04015908/Prot_SAP_000.pdf